CLINICAL TRIAL: NCT03028207
Title: New Study on the Prevalence of COPD in Spain EPI-Scan-II Study
Brief Title: A Cross-sectional Study on COPD Prevalence
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: IMS Health (Other)
Responsible Party: Sponsor
Other Study IDs: 205932
Record Dates: First submitted 2016-11-21; First posted 2017-01-23 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: EPI-Scan-II Study; COPD; Epidemiology; Spain; Chronic Obstructive Pulmonary Disease; Prevalence; Cross-sectional
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Subjects with FEV1/FVC score less than 0.70 post-bronchodilator test will be allocated to COPD group and the prevalence of COPD will be evaluated. Subjects in this group will be categorized in 4 groups namely GOLD I - IV depending on the disease severity.
  Interventions: Procedure: Medical tests; Other: Questionnaire
- Non-COPD: Subjects with FEV1/FVC score greater than or equal to 0.70 post-bronchodilator test will be allocated to non-COPD group.
  Interventions: Procedure: Medical tests; Other: Questionnaire

INTERVENTIONS:
Procedure: Medical tests — During Visit 1, subjects will go through medical tests including spirometry, bronchodilation test, pulse oximetry, cooximetry, and bioimpedance. Additional tests will be performed at up to 9 centers such as pulmonary diffusion test, 6 minute walk test, CT during the same visit.
Other: Questionnaire — During Visit 1, subjects will be given an Electronic Case Report Form (eCRF) with a series of questionnaire such as Health Related Quality of Life (HRQoL) CAT questionnaire, HADS anxiety scale, YPAS physical activity questionnaire, ECSC respiratory symptoms questionnaire, occupational exposure related questionnaire, MMSE questionnaire, Fagerstrom test, Prochaska test.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality worldwide and hence, estimating its prevalence is important. Since 2007, there are few data on the prevalence of COPD in the general population in Spain. The main objective of this epidemiological observational study is to estimate the prevalence of COPD in residents of Spain among the population over 40 years of age. The subjects will be distributed in two groups depending on the presence and absence of COPD. The study will have a single visit in which a brief interview will take place and subjects will need to complete the medical tests the case report form with a series of questionnaires. No drugs will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 40 years or older selected from the general population.
* Subjects who have provided oral consent to participate in the brief telephone interview; these subjects will need to sign the informed consent to continue participating in the study.

Exclusion Criteria:

* Subjects with any physical or cognitive difficulties which will prevent them from participating in any of the study tests (example, spirometry and questionnaires).
* Subjects who are not located, dead or displaced.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes individuals who, after the two telephone contacts, makes the study visit with the healthcare professional in the participating site and does not present any physical or cognitive difficulties that prevent conducting any of the study tests (e.g., spirometry, questionnaires).
Sampling Method: Probability Sample
Enrollment: 9362 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with COPD in Spain | Up to 9 months
  The prevalence of COPD in the subjects will be calculated according to the spirometric criteria, considering that a subject has COPD when the Forced Expiratory Volume in One Second/ Forced Vital Capacity (FEV1/FVC) obtained in post-bronchodilator spirometry is less than 0.7. The prevalence of COPD according to the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria will also be evaluated.

SECONDARY OUTCOMES:
Number of COPD exacerbations | Up to 9 months
  The No. and type of COPD exacerbations in the past year will be described. Depending on the frequency, the subjects will be grouped into two categories: less than two exacerbations per year and two or more exacerbations per year.
Analysis of differences in the prevalence of COPD and its evolution time | Up to 9 months
  Previous studies such as IBERPOC or EPISCAN will be analyzed to compare differences in the prevalence of COPD and its evolution over time.
Estimation of COPD prevalence by age and sex | Up to 9 months
  Subjects in COPD cohort will be classified according to sex and age groups, and the association between prevalence and age will be explored from the chi-squared test and linear-by-linear association. The prevalence of COPD in different age and sex groups will be compared according to the FEV1/FVC ratio.
Number of subjects with comorbidities | Up to 9 months
  Presence of comorbidities among subjects with and without COPD will be evaluated using the Charlson and COPD speciﬁc comorbidity test (COTE indices), which associate long-term mortality with subject comorbidity.
Evaluation of COPD severity among subjects using the GOLD severity classification | Up to 9 months
  COPD severity according to GOLD criteria will be evaluated from the results of FEV1/FVC from the post-bronchodilator test. Subjects will be classified into 4 groups namely GOLD 1, GOLD 2, GOLD 3 and GOLD 4 for COPD severity with GOLD 1= mild and GOLD 4 = very severe COPD.
Analysis of distribution of subjects according to Spanish COPD Guide (GesEPOC) | Up to 9 months
  Subjects will be distributed based on GesEPOC into 4 phenotypes that determine differential treatment: non-exacerbator; mixed COPD-asthma; exacerbator with emphysema and exacerbator with chronic bronchitis.
Analysis of the risk factors of COPD | Up to 9 months
  The risk factors of COPD including level of physical activity, degree of smoking, occupational exposure and exposure to smoke from biomass combustion will be analyzed in COPD cohort.
Assessment of relationship between the diagnosis of COPD, symptoms, level of physical activity and smoking status | Up to 9 months
  The relationship between the diagnosis of COPD, the level of physical activity and smoking will be assessed first by describing physical activity and smoking based on study cohorts. In the subpopulation of subjects who are smokers, the score on the Fagerstrom Test calculated as the sum of the 6 items (0-10) will be described and it will also be categorized as follows: mild dependency (0-2), medium dependency (3-5) and high dependency (6-10), as well as the smoking cessation phase in which they are, as assessed by Prochaska's stage: pre-contemplation, contemplation, preparation, action, maintenance, termination and relapse.
Assessment of treatment received according to current guideline | Up to 9 months
  It will be assessed whether treatment received in the study's COPD population complies with current regulations. The rate of undertreatment and overtreatment in subjects with COPD will also be evaluated. The percentage of COPD subjects who are treated according to the provisions of GesEPOC and according to GOLD will be compared in a post hoc analysis.
Number of subjects with smoking habit | Up to 9 months
  The prevalence of smoking and electronic cigarette use in people of 40 years of age or older in Spain and by sex will be described.
Degree of nicotine dependence among subjects | Up to 9 months
  The level of nicotine dependence among smokers will be assessed using Fagerstrom test. The test will consist of 6 items and the final score will range from 0- 10 with higher score correlating with higher nicotine dependency. The phase of smoking cessation of subjects will also be assessed using the Prochaska's test. In this test, 3 questions will be asked to each subject. It will identify the smoker's time of addiction to tobacco based on a series of set stages: pre-contemplation, contemplation, preparation, action and maintenance.
Number of subjects with respiratory symptoms | Up to 9 months
  The presence and prevalence of specific respiratory symptoms such as chronic cough, dyspnea will be estimated using the European Coal and Steel Community (ECSC) respiratory symptoms questionnaire. The questions will be divided into 6 sections namely cough, expectoration, dyspnea, wheezing and intra-thoracic pressure, asthma attacks and treatments.
To evaluate Health Related Quality of Life (HRQoL) of subjects | Up to 9 months
  HRQoL will be evaluated by using the COPD Assessment Test (CAT) questionnaire. It will consist of a single dimension with 8 items, each with a response scale of 0 (no limitation) to 5 (very limited). The items will assess the degree of severity of cough, presence of mucus, chest pressure, dyspnea, limited domestic activities, social limitations and limited sleep and energy. The overall score will be described in a range of 0-40 points and will distribute subjects into two groups including CAT less than 10 (low impact of COPD) and CAT more than or equal to 10 (medium/high impact of COPD on the subject).
Number of subjects with possible cognitive impairment | Up to 9 months
  Possible cognitive impairment will be evaluated in subjects 60 years of age or older using mini-mental state examination (MMSE) questionnaire. It is a rapid screening test for dementia and its evolutionary staging. The test consists of 30 items and will explore five cognitive areas: orientation, fixation, concentration and calculation, memory and language. The total score will range from 0 to 30 points. If the score falls between 0-22, the subject will be considered to have a cognitive deficit and those achieving score from 23-30 will be concluded as subjects without a cognitive deficit.
Number of subjects with anxiety/depression | Up to 9 months
  The presence of anxiety and depression among the subjects will be assessed using the Hospital Anxiety and Depression Scale (HADS). The HADS has two components that include scores for anxiety and depression. The response options are Likert-type, ranging from zero to three, giving a scoring range of 0-21 each. Depending on the HADS score, the subjects will be divided into 3 categories HADS 0-7 (absence of clinically relevant anxiety and/or depression), HADS 8-10 (likely to require consideration), HADS 11-21 (presence of anxiety/ depression relevant symptoms).
Evaluation of lean mass index among subjects | Up to 9 months
  The percentage of lean mass index will be evaluated and compared between COPD and non-COPD subjects by using bioimpedance. Body composition will be measured based on the electrical properties of biological tissues.
Evaluation of exercise tolerance among subjects | Up to 9 months
  Exercise tolerance between COPD and non-COPD subjects will be evaluated with the help of 6 minute walk test. The distance in meters and the reason for the stop will be measured, along with the initial and final heart rate and initial and final saturation of oxyhemoglobin (SatO2).
To evaluate daily physical activity of subjects | Up to 9 months
  The daily physical activity of COPD and non-COPD subjects will be compared using the Yale Physical Activity Survey (YPAS) questionnaire. YPAS will be calculated as the sum of the 5 sub-indices: index of vigorous activity, easy stroll index, moving index, standing index and sitting index. This index will range from 0 to 137 points. The subjects will be categorized into two groups namely YPAS less than 51 (sedentary subjects) and YPAS more than or equal to 51 (not sedentary subjects).
Recording of age | Up to 9 months
  Age will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in this study.
Number of subjects with different sociodemographic characteristics | Up to 9 months
  No. of subjects with different education level, gender, marital and smoking status will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in this study.
Recording of body mass index (BMI) | Up to 9 months
  BMI will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in this study.
Number of instances of underdiagnosis and overdiagnosis of COPD in subjects | Up to 9 months
  No. of instances of underdiagnosis will be described in the subsample of subjects who, despite declaring they had never received a previous diagnosis of COPD, reflect the presence of the disease from the study results. Also, the no. of instances of overdiagnosis will be described among those who claim having a prior diagnosis of COPD but who show this diagnosis to be unconfirmed after the study results. The correlation between the two variables will be analyzed using the Kappa index.
Number of subjects with abnormal multidimensional assessment of COPD | Up to 9 months
  No. of subjects with abnormal BMI, airflow Obstruction, Dyspnea and Exercise capacity (BODE) index ranging from 0-10 points and BMI, degree of dyspnea, pulmonary function and severe exacerbation (BODEX) index ranging from 0- 9 points will be recorded during multidimensional assessment of COPD.
Number of subjects with abnormal density of lung attenuation and thickness of airway caliber | Up to 9 months
  No. of subjects with attenuation of the lung parenchyma and thickness of the wall of the airway will be determined with the help of computed tomography (CT). No. of subjects with other abnormal parameters including the percentage of emphysema, extension areas, thickness of the airway, volume of the chest muscles, diameter of aorta vs. pulmonary artery, air trapping or coronary calcifications, bronchiectasis and fibrosis will also be assessed.
Number of subjects with dyspnea and other respiratory symptoms, health-related quality of life, exercise tolerance, physical activity and systemic inflammation among COPD and non-COPD subjects | Up to 9 months
  No. of subjects with intensity of dyspnea and other respiratory symptoms, health-related quality of life, exercise tolerance, physical activity and systemic inflammation will be assessed and compared between the COPD and non-COPD subjects depending on the amount of diffusion lung capacity.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Spain (20):
  - GSK Investigational Site, Avilés/Asturias
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Huesca
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pama de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo-Pontevedra
  - GSK Investigational Site, Vitoria-Gasteiz
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Rio F, Miravitlles M, Soriano JB, Cosio BG, Soler-Cataluna JJ, Casanova C, de Lucas P, Alfageme I, Rodriguez Gonzalez-Moro JM, Sanchez Herrero MG, Ancochea J; EPISCAN II study. Prevalence of reduced lung diffusing capacity and CT scan findings in smokers without airflow limitation: a population-based study. BMJ Open Respir Res. 2023 Jan;10(1):e001468. doi: 10.1136/bmjresp-2022-001468. PMID 36707127
- [Derived] Alfageme I, de Lucas P, Ancochea J, Miravitlles M, Soler-Cataluna JJ, Garcia-Rio F, Casanova C, Rodriguez Gonzalez-Moro JM, Cosio BG, Sanchez G, Soriano JB. 10 Years After EPISCAN: A New Study on the Prevalence of COPD in Spain -A Summary of the EPISCAN II Protocol. Arch Bronconeumol (Engl Ed). 2019 Jan;55(1):38-47. doi: 10.1016/j.arbres.2018.05.011. Epub 2018 Jul 7. English, Spanish. PMID 30612602